CLINICAL TRIAL: NCT03588871
Title: Comparison of the Efficacy and Quality of Life of Three Bleaching Products
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo de Investigação em Bioquímica e Biologia Oral (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL16001
Record Dates: First submitted 2018-05-04; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-05

CONDITIONS: Tooth Bleaching; Quality of Life
Keywords: Tooth bleaching; Quality of life
MeSH Terms: interventions — Vivastyle; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A (Experimental): Dental bleaching with PaintOn Plus, HP 6%, 6x10min, two sessions
  Interventions: Other: Dental bleaching with PaintOn Plus VivaStyle; Other: Dental Bleaching impact in quality of life with PaintOn Plus Vivastyle
- Group B (Experimental): Dental bleaching with Opalescence GO, HP 6%, 10x60min
  Interventions: Other: Dental bleaching with Opalescence GO; Other: Dental Bleaching impact in quality of life with Opalescence GO
- Group C (Experimental): Dental bleaching with Opalescence PF, CP 16%, 14x60h
  Interventions: Other: Dental bleaching with Opalescence PF; Other: Dental Bleaching impact in quality of life with Opalescence PF

INTERVENTIONS:
Other: Dental bleaching with PaintOn Plus VivaStyle — Procedure of tooth bleaching using products with 6% hydrogen peroxide or its equivalent, specifically the PaintOn Plus Vivastyle 6% HP (Ivoclar Vivadent)
  Arms: Group A
Other: Dental Bleaching impact in quality of life with PaintOn Plus Vivastyle — Evaluation of oral quality of life after dental bleaching treatment with PaintOn Plus Vivastyle 6% HP (Ivoclar Vivadent) using an oral quality of life measuring questionnaire, specifically the Oral Health Impact Profile-14
  Arms: Group A
Other: Dental bleaching with Opalescence GO — Procedure of tooth bleaching using products with 6% hydrogen peroxide or its equivalent, specifically the Opalescence GO 6% HP (Ultradent)
  Arms: Group B
Other: Dental Bleaching impact in quality of life with Opalescence GO — Evaluation of oral quality of life after dental bleaching treatment with Opalescence GO 6% HP (Ultradent) using an oral quality of life measuring questionnaire, specifically the Oral Health Impact Profile-14
  Arms: Group B
Other: Dental bleaching with Opalescence PF — Procedure of tooth bleaching using products with 6% hydrogen peroxide or its equivalent, specifically the Opalescence PF 16% CP (Ultradent)
  Arms: Group C
Other: Dental Bleaching impact in quality of life with Opalescence PF — Evaluation of oral quality of life after dental bleaching treatment with Opalescence PF 16% CP (Ultradent) using an oral quality of life measuring questionnaire, specifically the Oral Health Impact Profile-14
  Arms: Group C

SUMMARY:
The aims of this study are: to compare the efficacy of three different dental bleaching products; to evaluate colour relapse following dental bleaching treatment at 1, 3 and 6 months follow up; to evaluate the impact in quality of life from dental bleaching treatments.

Products to be used represent three different techniques and formulations: in office, universal tray and custom tray (respectively VivaStyle Paint On Plus (Ivoclar Vivadent, Liechtenstein), Opalescence GO 6% (Ultradent, USA) and Opalescence PF 15% (Ultradent, USA).

All products contain 6% hydrogen peroxide or its equivalent.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Be willing to refrain from use of tobacco products during the study
* Be willing to sign an informed consent form
* At least one teeth 13,11,21,23,33,43 has a gradable VITA shade A3,5 or darker by clinical assessment

Exclusion Criteria:

* Teeht with restorations in frontal teeth
* Patients with untreated periodontitis or caries
* Patients with fixed orthodontics appliances
* Patients with know allergies to ingredients
* Patients who are nursing or pregnant
* Patients with severe systemic illnesses
* Patients with development tooth anomalies
* Patients with non vital anterior teeth
* Patients with insufficient oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Change on visually determination of tooth colour | 2 weeks (before and after treatment)
  Determination of tooth colour using a visual tooth shade guide
Change on spectrophotometer determination of tooth colour | 2 weeks (before and after treatment)
  Determination of tooth colour using a spectrophotometer
Subjective evaluation of tooth colour change during follow-up | 1, 3 and 6 months
  Determination of tooth colour relapse using visual tooth shade guide (VITA shade guide)
Change on quality of life during treatment and follow-up | 2 weeks (before and after treatment), 1 month, 3 months and 6 months
  Impact on quality of life using an oral quality of life measuring questionnaire, the Oral Health Impact Profile 14 (OHIP-14). The OHIP-14 ranges from 0 to 56 (final sum of all the seven subscales), with higher scores indicating poorer quality of life.
Objective evaluation of tooth colour change during follow-up | 1, 3 and 6 months
  Determination of tooth colour relapse using a spectrophotometer

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine of the University of Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No